CLINICAL TRIAL: NCT00051779
Title: A 24-Week Blinded Study Conducted at Multiple Centers, Evaluating the Safety and Effectiveness of Various Doses of the Investigational Drug (CAL) Versus Zoledronic Acid (Zometa®) When Randomly Assigned to Patients With Breast Cancer That Has Metastasized to Bone
Brief Title: An Investigational Drug (CAL) Versus Zoledronic Acid (Zometa®) in Patients With Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chugai Pharma USA (Industry)
Purpose: Treatment
Other Study IDs: CAL-03
Record Dates: First submitted 2003-01-16; First posted 2003-01-17 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-02

CONDITIONS: Breast Neoplasms; Breast Cancer; Metastasis
Keywords: CAL; Parathyroid hormone-related protein (PTHrP); Breast Cancer; Bone Metastasis; Hypercalcemia
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Hypercalcemia

INTERVENTIONS:
Drug: CAL

SUMMARY:
This study is intended to evaluate the safety, tolerability, and possible effectiveness of an investigational humanized monoclonal antibody (CAL) to the parathyroid hormone-related protein (PTHrP) when compared to zoledronic acid in patients with breast cancer metastatic to bone.

The study will also evaluate the possible effects of both study drugs on performance status, markers of bone metabolism, and skeletal events related to bone metastasis including elevated blood calcium levels, bone pain, metastatic lesions, complications and interventions. The levels of CAL in the blood will also be evaluated.

ELIGIBILITY:
Major Inclusion Criteria - Others Stipulated within the Protocol

The study physician must assure you have/are:

* Must be a female at least 18 years of age and be using an effective form of birth control.
* A documented history of breast cancer and at least one bone metastasis that has not been previously treated by radiation or surgery, and is not anticipated to be treated within the next 24 weeks.
* A total body bone scan and other radiographic scan(s) performed on you within 4 weeks prior to or during the screening period sufficient to image all sites of bone metastases.
* You must be willing to perform a daily telephone diary and be willing to keep a paper diary and provide voluntary consent to participate in this study.

Major Exclusion Criteria - Others Stipulated within the Protocol

The study physician must assure you do not have/are not:

* A change in analgesic (pain relief) type medication during the screening period (example, non-narcotic to narcotic).
* Received radiation therapy to any bone metastasis or started a new course of chemotherapy within 3 weeks prior to the screening visit or during the screening period.
* Used any bisphosphonate type drug during the 30 days prior to the anticipated first dose of study drug
* Vertebral spine or weight-bearing bone metastasis that would place you at imminent risk for fracture or surgical intervention.
* Evidence of active infection or immune deficiency, renal failure, abnormal liver function, or a serum calcium level > 10.1 mg/dL.
* Use of any investigational drug within 30 days prior to screening.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (38):
- United States (38):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Bay Area Cancer Research Group, Concord, California
  - California Cancer Care, Inc., Greenbrae, California
  - Institute of Cancer Therapies, Los Angeles, California
  - San Diego Cancer Research Institute, Vista, California
  - Anschutz Cancer Pavilion at the University of Colorado Cancer Center, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Rush Cancer Institute, Chicago, Illinois
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Louisiana State University, New Orleans, Louisiana
  - Frederick Memorial Hospital, Frederick, Maryland
  - Dana-Farber/Harvard Cancer Center, Boston, Massachusetts
  - Josephine Ford Cancer Center, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Southfield Oncology Institute, Inc., Southfield, Michigan
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - Nevada Cancer Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - HemOnCare, P.C., Brooklyn, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ireland Cancer Center, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Hematology Oncology Consultants, Inc., Columbus, Ohio
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Palmetto Health, Columbia, South Carolina
  - Boston Baskin Cancer Group, Memphis, Tennessee
  - The Boston Baskin Cancer Group, Memphis, Tennessee
  - The West Clinic, Memphis, Tennessee
  - Cancer Specialists of South Texas, PA, Corpus Christi, Texas
  - Center for Oncology Research & Treatment, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Medical College of Wisconsin-FMLH East Neoplastic Diseases and Related Disorders, Milwaukee, Wisconsin